CLINICAL TRIAL: NCT01047891
Title: A Randomized, Double-blind, Placebo Controlled, Multicenter Phase II Study to Assess the Efficacy and Safety of Sorafenib Added to Standard Treatment With Topotecan in Patients With Platinum-resistant Recurrent Ovarian Cancer
Brief Title: Efficacy and Safety Study of Sorafenib With Topotecan in Patients With Platinum-resistant Recurrent Ovarian Cancer
Acronym: TRIAS 2009
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JSehouli (Other)
Responsible Party: Sponsor-Investigator, JSehouli, Prof. Dr. med, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRIAS 2009
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Topotecan 1,25 mg/m²/d administered as an i.v. infusion over 30 minutes once daily on days 1-5, every 21 days and Sorafenib 400 mg orally twice daily (total daily dose 800 mg) administered
  Other Names: Nexavar®

SUMMARY:
It is assumed, that the patients of the standard arm show a median progression-free survival time of 4.4 months those of the experimental arm of at least 6.9 months. Assuming a recruitment period of 18 months and follow-up for at least 12 months a total sample size of 174 patients is required (two-sided, α=0.05, 80% power). To account for 5% drop-outs 184 patients will be randomized.

A Data Monitoring and Safety Board (DMSB) will be established. This board will evaluate the safety profile of the drug combination after 6 patients and after 12 patients have received 1 cycle of treatment.

DETAILED DESCRIPTION:
Ovarian cancer continues to be a leading cause of cancer-related deaths in women and is the leading cause of deaths attributed to gynecologic malignancies. Because ovarian cancer is usually asymptomatic in its early stages, the disease often has spread outside of the pelvic region at the time of diagnosis and requires debulking surgery followed by systemic chemotherapy. First-line chemotherapy involves platinum-based treatments, including the widely adopted regimens of cisplatin/paclitaxel, carboplatin/paclitaxel, and single-agent carboplatin. Although these regimens yield relatively satisfactory tumor response rates, the majority of patients experience disease recurrence and receive additional treatments. For such patients, a number of antitumor agents with novel mechanisms of action (topotecan, gemcitabine, pegylated liposomal doxorubicin, docetaxel, etoposide) have been applied, in addition to retreatment with platinum, with the goal of re-establishing remission or disease control, minimizing disease-related symptoms, improving quality of life, and extending patient survival. Of these agents, topotecan (Hycamtin®; GlaxoSmithKline) is one of the best-characterized agents in the recurrent setting.

Topotecan is an S-phase 1-dependent cytotoxic agent that targets the topoisomerase I enzyme and exhibits broad activity in solid tumors and is approved for the treatment of recurrent ovarian cancer in US and in most western countries.

Data from preclinical and clinical studies reported in the last 2 years demonstrate the importance of several proangiogenic factors in the tumorigenesis and prognosis of ovarian cancer, suggesting possible new targets for antiangiogenic therapy. Once-daily oral treatment with Sorafenib produces broad spectrum antitumor efficacy in preclinical tumor models including also xenograft models of ovarian carcinoma. Preliminary antitumor activity has been reported in single ovarian cancer patients in several phase I and phase II studies.

Most promising strategy in the therapy of advanced and recurrent ovarian cancer seems to be the combination of cytotoxic agents and targeted therapies. Furthermore an oral therapy to achieve and maintain long term tumor control seems to be very attractive.

Therefore Sorafenib and Topotecan would make a rational therapeutic strategy for combination in recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed epithelial ovarian cancer, primary peritoneal carcinomatosis or fallopian tube cancer
2. Patients must have platinum resistant (relapse-free interval < 6 months of a platinum-containing primary or secondary therapy) or platinum refractory (progression during primary or secondary platinum treatment) disease defined by measurable disease according to RECIST or elevated CA-125 level according the GCIG-criteria.

   Definition of relapse: Demonstration of measurable or non-measurable tumour according to RECIST criteria by an imaging procedure (where applicable before relapse surgery) or increase in the tumour marker CA-125 to twice the upper laboratory value of normal for the hospital or histological confirmation of tumour relapse by biopsy or surgery.
3. No more than 2 prior treatment regimens for recurrent epithelial ovarian cancer.
4. Elevated CA-125-value before study entry in order to assess the response according the GCIG-criteria (see below). Patients without elevated CA-125 may be enrolled if they show a measurable or not-measurable disease (according RECIST) evaluated by imaging techniques (measurable disease - at least one unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan) or histologically or cytologically confirmed relapse
5. ECOG Performance Status of 0 or 1
6. ≥ 18 years age
7. The patient must be recovered from a prior operation. The operation must be performed at least 4 weeks prior to start of study drug,
8. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening

   * Hemoglobin ≥ 9.0 g/dl
   * Leucocyte count ≥ 3.000/micro liter
   * Absolute neutrophil count (ANC) major than 1.500/micro liter
   * Platelet count ≥ 100.000/micro liter
   * PT-INR/PTT < 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists].
   * Total bilirubin < 1,0 times the upper limit of normal
   * ALT and AST < 2,5 x upper limit of normal (< 5 x upper limit of normal for patients with liver involvement of their cancer); Alkaline phosphatase < 4 x ULN
   * Calculated creatinine clearance ≥ 50 ml/min or serum creatinine ≤ 1,2 x upper limit of institutional values (according to Cockcroft and Gault)
9. Life expectancy of at least 12 weeks
10. Signed and dated written informed consent before the start of specific protocol procedures.

Exclusion Criteria:

1. History of cardiac disease: congestive heart failure >NYHA class 2; active coronary artery disease (CAD) or myocardial infarction within the past 6 months (MI more than 6 months prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled arterial hypertension with systolic blood pressure >160 mmHg or diastolic blood pressure > 90 mm Hg despite optimal treatment
2. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 5 years prior to study entry
3. Prior radiological or clinical evidence of CNS metastases including previously treated, resected, or asymptomatic brain lesions or leptomeningeal involvement by head CT scan or MRI
4. Known or suspected hypersensitivity reaction to topotecan or any ingredient of topotecan or sorafenib or any ingredient of sorafenib
5. Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
6. History of HIV infection or chronic hepatitis B or C
7. History of organ allograft
8. Patients with history of colon perforation
9. Patients with history of colitis or neutropenia colitis
10. Patients with evidence or history of bleeding diathesis
11. Serious non healing wound, fracture or ulcer
12. Patients undergoing renal dialysis
13. Patients unable to swallow oral medications
14. Significant disease which, in the investigator's opinion, would exclude the patient from the study
15. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
16. Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
17. Medical or psychological conditions that would not permit the subject to complete the study or sign informed consent
18. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
19. Legal incapacity or limited legal capacity
20. Participation in another clinical study with experimental therapy within the 30 days before start of treatment
21. Subjects housed in an institution on official or legal orders.

    Excluded therapies and medications, previous and concomitant:
22. Patients with prior therapy containing topotecan
23. Patients with prior therapy containing Avastin or other VEGFR TK1
24. Any other anticancer chemotherapy or immunotherapy or investigational drug therapy outside of this trial during the study or within 4 weeks prior to study entry.
25. Radiotherapy during study or within 4 weeks prior to start of study drug and prior radiotherapy of > 25% of the bone marrow (exception: palliative radiotherapy of non-target lesions or pain therapy or local bone irradiation)
26. Autologous bone marrow transplant or stem cell rescue within 4 months of study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2010-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Primary objective: Determination of the progression-free survival (PFS) of patients treated with topotecan and sorafenib versus topotecan and placebo | 18 months
  The primary target value of this study is the comparison of the median progression-free survival time between the two study arms. Progression-free survival time (PFS) of a patient is defined as the time in months from start of the first therapy cycle until PD or death is observed

SECONDARY OUTCOMES:
Overall survival | 18 months
  Overall survival (OS) of a patient being defined as the time in months from start of the first therapy cycle to death or the end of study
Response rate | 18 months
  Response rates, i.e. percentage of patients showing overall response (CR+PR), progression or stable disease
Duration of response | 18 months
  Duration of response is the time in months from first assessment of CR or PR until the first date of PD or death
Time to progression (TTP) | 18 months
  Time to progression (TTP) of a patient being defined as the time in months from start of the first therapy cycle until PD is observed
Safety and tolerability | 18 months
  Incidence and type of AE in terms of:
  * All AE,
  * Related AE,
  * SAE,
  * Related SAE,
  * NCI-CTC grade 3 and 4 AE,
  * Related NCI-CTC grade 3 and 4 AE,
  * AE leading to treatment discontinuation,
  * Incidence of, and reason for, deaths
Assessment of quality of life over time as defined by EORTC-QLQ C 30 and Ovar 28 questionnaire | 18 months
  Assessment of Quality of life over time as defined by EORTC-QLQ C 30 and Ovar 28 questionnaire and, in case of participation in the sub-study, FOSI questionnaire, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Jalid Sehouli Sehouli, Professor, Principal Investigator — Charité Campus Virchow-Klinikum, Berlin
Locations (1):
- Charité Campus Virchow-Klinikum, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Chekerov R, Hilpert F, Mahner S, El-Balat A, Harter P, De Gregorio N, Fridrich C, Markmann S, Potenberg J, Lorenz R, Oskay-Oezcelik G, Schmidt M, Krabisch P, Lueck HJ, Richter R, Braicu EI, du Bois A, Sehouli J; NOGGO; AGO TRIAS Investigators. Sorafenib plus topotecan versus placebo plus topotecan for platinum-resistant ovarian cancer (TRIAS): a multicentre, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Oncol. 2018 Sep;19(9):1247-1258. doi: 10.1016/S1470-2045(18)30372-3. Epub 2018 Aug 9. PMID 30100379